CLINICAL TRIAL: NCT04791475
Title: Comparison Of Dexmedetomidine And Dexamethasone As An Adjuvant To Bupivacaine In Ultrasound Guided Supraclavicular Brachial Plexus Block In Upper Limb Surgeries
Brief Title: Comparison Of Dexmedetomidine And Dexamethasone As An Adjuvant To Bupivacaine In Brachial Plexus Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Principal Investigator, manu bhattarai, Dr. Manu Bhattarai, Resident, Tribhuvan University Teaching Hospital, Institute Of Medicine.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TribhuvanUTH
Record Dates: First submitted 2021-03-05; First posted 2021-03-10 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Brachial Plexus Block; Dexmedetomidine; Dexamethasone; Bupivacaine
Keywords: Brachial Plexus Block; Dexmedetomidine; Dexamethasone; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine with 0.5% bupivacaine (Experimental): 1mcg/kg dexmedetomidine as an adjuvant to 0.5% bupivacaine 20 ml in USG guided Supraclavicular Brachial Plexus Block
  Interventions: Procedure: adding Dexmedetomidine and dexamethasone to bupivacaine in USG guided supraclavicular brachial plexus block.
- Dexamethasone with 0.5% bupivacaine (Active Comparator): 4mg dexamethasone as an adjuvant to 0.5% bupivacaine 20 ml in USG guided Supraclavicular Brachial Plexus Block
  Interventions: Procedure: adding Dexmedetomidine and dexamethasone to bupivacaine in USG guided supraclavicular brachial plexus block.

INTERVENTIONS:
Procedure: adding Dexmedetomidine and dexamethasone to bupivacaine in USG guided supraclavicular brachial plexus block. — The linear transducer probe (frequency 4 -12 Hz) of USG machine will be used. A superficial skin wheal will be made by 2ml of 1% lignocaine subcutaneously at the point of needle insertion. USG guided Brachial plexus block will be performed by supraclavicular route via the subclavian perivascular approach in in-plane technique from lateral to medial using 22 gauge spinal needle. Study Drug will be administered via Pressure Monitoring line connected to syringe according to the allocated group with repeated aspiration and incremental dosing. • Intercostobrachial nerve block will be performed to alleviate the tourniquet pain. A 25 G needle will be inserted at the level of axillary fossa. The entire width of the medial aspect of arm, starting at the deltoid prominence and proceeding inferiorly, will be infiltrated with 5ml of 1% Lignocaine with Epinephrine (1:4,00,000) to raise a subcutaneous wheal. •

SUMMARY:
Brachial plexus block is a regional anaesthesia technique employed as a safe and valuable alternative to general anaesthesia for upper limb surgery. In recent practices of day care surgeries, brachial plexus block seems to be a better alternative to general anesthesia with minimal hospital stay and better analgesic effect. Among several techniques of brachial plexus block, supraclavicular approach is considered as easiest, effective and can be performed much more quickly than other approaches. Various local anaesthetic agents and adjuvants are used for this purpose. Among them, bupivacaine has been the most widely used long-acting local anaesthetic agent. Combining local anesthetics with different adjuncts can prolong the duration of analgesia associated with brachial plexus block. Among various adjuncts, dexamethasone and dexmedetomidine have been identified as clinically effective adjuncts. Several metaanalyses have convincingly demonstrated their efficacy in prolonging the analgesic duration of brachial plexus block. However, there has been limited research conducted to compare the effects of dexamethasone and dexmedetomidine added as adjuvants to the local anesthetics for BPB. Studies have demonstrated benefits of one agent over other without any definitive conclusion as which is the best agent for this purpose. Therefore, there is a need of study to compare the onset and duration of bupivacaine when dexmedetomidine or dexamethasone is used as an adjuvant to bupivacaine for ultrasound-guided supraclavicular BPB

DETAILED DESCRIPTION:
Peripheral nerve block (PNB), as an integral part of regional anesthetic technique, remains a well-accepted component of comprehensive anaesthetic care. William Halstead (1852-1922) was first to perform Brachial Plexus Block (BPB) in 1884 by surgically exposing the roots of the brachial plexus and injecting each nerve directly. Kulenkampff described the first percutaneous supraclavicular approach in 1911. BPB provides both intraoperative anaesthesia as well as postoperative analgesia. Being a regional anaesthetic technique, it has many advantages over general anaesthesia like effective analgesia with good motor blockade, awake patient, extended postoperative analgesia, early mobilization, no airway manipulation, avoidance of polypharmacy and decreased incidence of postoperative nausea and vomiting. Advantages of supraclavicular approach include rapid onset and reliable blockade with a small volume of local anaesthetic and produced a more intense motor blockade and reduced the incidence of Horner's syndrome compared with Interscalene BPB. The clinical indications of supraclavicular BPB have been confined to upper limb surgeries below the midshaft of humerus because of concerns that it is performed too distally from the cervical nerve roots to block the suprascapular nerve which innervates 70% of the shoulder joint in addition to the subacromial bursa, coracoclavicular ligament, and acromioclavicular joint. There is evidence that peripheral nerve blocks performed by ultrasound guidance alone, or in combination with Peripheral Nerve Stimulator (PNS), are superior in terms of improved sensory and motor block, reduced need for supplementation and fewer minor complications reported. Using ultrasound alone shortens performance time when compared with nerve stimulation, but when used in combination with PNS it increases performance time. Many local anaesthetics have been used to produce brachial plexus block. Most common among them is bupivacaine, because of its higher potency and prolonged duration of action. Bupivacaine is an amide local anaesthetic. It prevents transmission of nerve impulses by inhibiting passage of sodium ions through selective ion channel in nerve membranes. This slows the rate of depolarization such that threshold potential is not reached and action potential not propagated. The half life of bupivacaine in adults is 3.5 hours. The commonly used concentrations in brachial plexus block are 0.25%, 0.375% and 0.5%. Studies have shown that mass of bupivacaine rather than concentration is the major determinant of the Effective Dose 50 (ED50) for achieving supraclavicular brachial plexus block. The concentration of bupivacaine that will be used in our study is 0.5% and volume is 20 ml. Adjuvants or additives are often used with local anaesthetics for its synergistic effect by prolonging the duration of sensory-motor block and limiting its cumulative dose requirement. Various drugs like opioids, epinephrine, alpha-2 adrenergic antagonists, steroids, anti-inflammatory drugs, midazolam, ketamine, magnesium sulfate and neostigmine have been used to potentiate the effect of local anesthetics. Due to its potential adverse effects, current researches are exploring newer drugs and delivery mechanisms to prolong the duration of action of local anesthetics. Recently, dexamethasone and dexmedetomidine have been identified as clinically effective adjuncts; several metaanalyses have convincingly demonstrated their efficacy and prolonging the analgesic duration of PNB. Dexmedetomidine, a potent α2 adrenoceptor agonist, is approximately eight-times more selective towards the α2 adrenoceptor than clonidine. Dexmedetomidine is also reportedly safe and effective when administered with long-acting local anesthetics in PNBs. No significant histopathologic abnormalities were reported after intrathecal or perineural administration of dexmedetomidine. There have been four proposed mechanisms for the action of alpha 2 adrenergic agonists in peripheral nerve blocks. These mechanisms include centrally mediated analgesia, ∝2B-adrenoceptor mediated vasoconstrictive effects, attenuation of the inflammatory response, and direct action on the peripheral nerve. In this study we are adding 1mcg/kg dexmedetomidine as adjunct to bupivacaine as previous studies have shown that 1 mcg/kg dexmedetomidine added perineurally to levobupivacaine in Supraclavicular BPB is a safer dose than 2 mcg/kg with less sedation, bradycardia, and comparable analgesia. Dexamethasone is a very potent and highly selective glucocorticoid. Various studies have been done using dexamethasone as an adjuvant to local anaesthetics mixture in brachial plexus block resulting in variable effects on onset but prolonged duration of analgesia and motor block. Dexamethasone produces analgesia by blocking pain signal transmission in nociceptive c-fibers, suppressing ectopic neural discharge and by inhibiting the action of phospholipase A2. The block prolonging effect of peripherally applied dexamethasone could be due to alteration in the function of potassium channels in the excitable cells by dexamethasone via glucocorticoid receptors present in the brachial plexus. It may also be due to the local vasoconstrictive effect of dexamethasone via glucocorticoid receptors. In this study we are using 4 mg dexamethasone as articles have shown that perineural dexamethasone at a dose of 4 mg prolongs the duration of analgesia after local anaesthetic PNB with efficacy similar to a dose of 8 mg and without any reported serious adverse effects. However, each of these molecules is associated with undesirable side effects: increased glycemia, neurotoxicity and risk of precipitation may occur after use of dexamethasone but studies show that these toxicities are very unlikely with peripheral use and at the low dose of 4mg which will be used in this study; bradycardia, hypotension, and sedation for dexmedetomidine. Importantly, most published trials of dexamethasone and dexmedetomidine have compared these adjuncts to control, with very scant head-to-head comparison. Notably, literature is characterized by conflicting results and inconsistent reporting of side effects.

ELIGIBILITY:
Inclusion Criteria:

* ASA PS I & II
* Age: 18-65 years
* Sex: Both male and female
* Patients scheduled for Upper limb surgery below the level of midshaft of humerus

Exclusion Criteria:

1. Local infection at the site of puncture
2. Patients having any neurologic deficit in the upper limb
3. Pregnant or lactating women.
4. Patients receiving adrenoceptor agonist or antagonist therapy or chronic analgesic therapy.
5. Patients with diabetic neuropathy, peripheral vascular disease, coagulopathy, or known allergies.
6. Patients with polytrauma.
7. Patients weighing <30 kg and > 100 kg.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
duration of analgesia | 20 hours
  The time between drug administration and request for first analgesic medication or NRS (numerical rating scale) score more than or equal to 4 will be recorded as duration of analgesia

SECONDARY OUTCOMES:
onset and duration of sensory blockade | 20 hrs
  The extent of sensory blockade will be tested in the median, radial, ulnar, and musculocutaneous nerve distribution using pinprick: 0 = no perception, 1 = decreased sensation, or 2 = normal sensation. • Successful blockade will be defined as complete sensory blockade (ie, sensory block score = 0) in the distribution of the radial, ulnar, median, and musculocutaneous nerves within 30 mins of performing the BPB.
onset and duration of motor blockade | 20 hrs
  Motor blockade assessment will be done using the modified Bromage scale for upper extremities on a three-point scale: Grade 0 : Normal motor function with full flexion and extension of elbow, wrist, and fingers Grade 1 : Decreased motor strength with ability to move the fingers only Grade 2 : Complete motor block with inability to move fingers • Motor blockade will be evaluated every 5 mins after injection of study drug for 30 mins or until complete motor block is achieved, whichever is earlier. • Onset time of motor block is defined as minimum of grade 1 of Modified Bromage scale
To assess for adverse events | 20 hrs
  bradycardia and hypotension , sedation, nausea vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Manu Bhattarai, Principal Investigator — MD resident
Locations (1):
- Tribhuvan University Teaching Hospital, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vorobeichik L, Brull R, Abdallah FW. Evidence basis for using perineural dexmedetomidine to enhance the quality of brachial plexus nerve blocks: a systematic review and meta-analysis of randomized controlled trials. Br J Anaesth. 2017 Feb;118(2):167-181. doi: 10.1093/bja/aew411. PMID 28100520